CLINICAL TRIAL: NCT02703779
Title: An Exploratory Trial to Estimate the Proportion of Patients With Tumor Cell Contaminated, Flow Positive Leukapheresis Products Collected With and Without Bortezomib as In-vivo Purging Prior to Autologous Stem Cell Harvest for Multiple Myeloma
Brief Title: Exploratory Trial to Estimate Proportion of Patients With Tumor Cell Contaminated Leukapheresis Products With and Without Bortezomib With In-vivo Purging - Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Siddhartha Ganguly (Other)
Responsible Party: Sponsor-Investigator, Siddhartha Ganguly, Medical Doctor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-IIT-BMT-MM-AutoSCT
Record Dates: First submitted 2016-02-18; First posted 2016-03-09 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Autologous; Stem Cell; Purging; In-vivo purging; Ex-vivo purging; Leukapheresis; Contaminated; Stem Cell Harvest; Stem Cell Transplant; Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Granulocyte Colony-Stimulating Factor; Filgrastim; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem cell collection without in-vivo purging with Bortezomib (Active Comparator): Standard of Care Stem cell collection without in-vivo purging with Bortezomib. Standard of Care drugs Granulocyte colony-stimulating factor (G-CSF) +/- Mozobil (the latter if needed).
  NOTE: Multiparametric Flow Cytometry to be performed on samples for BOTH groups A and B
  Interventions: Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Mozobil
- Stem cell collection with in-vivo purging with Bortezomib (Experimental): Bortezomib will be given subcutaneously (SQ) at 1.3 mg/m2 on day -11 and day -8 followed by Granulocyte colony-stimulating factor (G-CSF) given SQ on day -4 thru day -1 and continued until the collection is completed. Mozobil will be given if needed.
  There must be at least 72 hours between each dose of bortezomib. NOTE: Multiparametric Flow Cytometry to be performed on samples for BOTH groups A and B
  Interventions: Drug: Bortezomib; Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Mozobil

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be given to Group B participants by injection under the skin 11 days and 8 days before stem cell collection.
  Other Names: VELCADE
  Arms: Stem cell collection with in-vivo purging with Bortezomib
Drug: Granulocyte colony-stimulating factor (G-CSF) — Granulocyte colony-stimulating factor (G-CSF) will be given to all participants by injection under the skin 4 days and 1 day before stem cell collection, and then continued until the stem cell collection is completed.
  Other Names: NEUPOGEN; filgrastim; filgrastim-sndz; Zarxio
Drug: Mozobil — Mozobil will be given to all participants by injection under the skin only if needed per Investigator.
  Other Names: plerixafor

SUMMARY:
Explore stem cell collection with or without bortezomib with in-vivo purging in multiple myeloma.

DETAILED DESCRIPTION:
High dose chemotherapy with autologous stem cell transplant has resulted in improved overall survival and is currently considered an effective first line therapy applicable to the majority of patients with multiple myeloma. However disease relapse is inevitable and remains the primary cause of mortality in this cohort.

The purpose of this study is to estimate the proportion of subjects with plasma cell contamination of harvested stem cell product in standard and treatment arms. The study will explore whether or not in-vivo purging of malignant tumor plasma cells will improve progression free survival (PFS) for patients.

The study will consist of two groups:

Group A: Standard of Care (SOC) stem cell collection without in-vivo purging with bortezomib. Granulocyte colony-stimulating factor (G-CSF) and Mozobil used if needed.

Group B: Bortezomib 1.3mg/m^2 will be given subcutaneously (SQ) on days -11 and -8 followed by Granulocyte colony-stimulating factor (G-CSF) on days -4 through -1 prior to stem cell harvest (day 0).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the inclusion criteria to participate in this study.
* Ability to understand, and the willingness to sign a written Informed Consent Form
* Diagnosis of multiple myeloma undergoing planned autologous stem cell transplantation
* Age ≥ 18 years
* Karnofsky Performance Status (KPS) 70 or above, Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2
* Adequate organ and marrow function as defined below:

  * leukocytes ≥ 3,000/micro Liter (mcL)
  * absolute neutrophil count ≥ 1,500/mcL
  * platelets ≥ 100,000/mcL
  * total bilirubin within normal institutional limits NOTE: For this study, subjects with bilirubin levels > 1.5 Upper Limit of Normal (ULN) are excluded from enrollment in this study.
  * Aspartate Aminotransferase (AST) ( Serum Glutamic Oxaloacetic Transaminase [SGOT]) ≤ 2.5 X institutional upper limit of normal
  * Alanine Aminotransferase (ALT) (Serum Pyruvic Glutamic Transaminase [SPGT]) ≤ 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy. Should a woman or partner become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and the investigator immediately.
* A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

Exclusion Criteria:

* Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.
* Current or anticipated use of other investigational agents. NOTE the following clarification for this study: Prohibited Concurrent Therapy:

Participation in clinical trials with other investigational agents that are not included in this trial, within 14 days of the start of this trial until 2 weeks after participant has received the last dose of bortezomib for mobilization.

* Hypersensitivity to bortezomib, boron or mannitol or Granulocyte colony-stimulating factor (G-CSF)
* Subject has received > 6 months of lenalidomide (Revlimid®) therapy prior to stem cell collection
* Subject has known brain metastases. Presence of brain metastases should be excluded from this clinical trial because of poor prognosis and because patients often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Grade 3 or higher peripheral neuropathy
* Bilirubin levels > 1.5 ULN
* Uncontrolled inter-current illness including, but not limited to

  * ongoing or active infection
  * symptomatic congestive heart failure
  * unstable angina pectoris
  * cardiac arrhythmia
  * psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing: There is a potential for congenital abnormalities and for this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha Ganguly, MD, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- The University of Kansas Medical Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawstron AC, Orfao A, Beksac M, Bezdickova L, Brooimans RA, Bumbea H, Dalva K, Fuhler G, Gratama J, Hose D, Kovarova L, Lioznov M, Mateo G, Morilla R, Mylin AK, Omede P, Pellat-Deceunynck C, Perez Andres M, Petrucci M, Ruggeri M, Rymkiewicz G, Schmitz A, Schreder M, Seynaeve C, Spacek M, de Tute RM, Van Valckenborgh E, Weston-Bell N, Owen RG, San Miguel JF, Sonneveld P, Johnsen HE; European Myeloma Network. Report of the European Myeloma Network on multiparametric flow cytometry in multiple myeloma and related disorders. Haematologica. 2008 Mar;93(3):431-8. doi: 10.3324/haematol.11080. Epub 2008 Feb 11. PMID 18268286

RESULTS

PARTICIPANT FLOW:
Groups:
- Stem Cell Collection Without In-vivo Purging With Bortezomib: Standard of Care Stem cell collection without in-vivo purging with Bortezomib. Standard of Care drugs Granulocyte colony-stimulating factor (G-CSF) +/- Mozobil (the latter if needed).
  NOTE: Multiparametric Flow Cytometry to be performed on samples for BOTH groups A and B
  Granulocyte colony-stimulating factor (G-CSF): Granulocyte colony-stimulating factor (G-CSF) will be given to all participants by injection under the skin 4 days and 1 day before stem cell collection, and then continued until the stem cell collection is completed.
  Mozobil: Mozobil will be given to all participants by injection under the skin only if needed per Investigator.
- Stem Cell Collection With In-vivo Purging With Bortezomib: Bortezomib will be given subcutaneously (SQ) at 1.3 mg/m2 on day -11 and day -8 followed by Granulocyte colony-stimulating factor (G-CSF) given SQ on day -4 thru day -1 and continued until the collection is completed. Mozobil will be given if needed.
  There must be at least 72 hours between each dose of bortezomib. NOTE: Multiparametric Flow Cytometry to be performed on samples for BOTH groups A and B
  Bortezomib: Bortezomib will be given to Group B participants by injection under the skin 11 days and 8 days before stem cell collection.
  Granulocyte colony-stimulating factor (G-CSF): Granulocyte colony-stimulating factor (G-CSF) will be given to all participants by injection under the skin 4 days and 1 day before stem cell collection, and then continued until the stem cell collection is completed.
  Mozobil: Mozobil will be given to all participants by injection under the skin only if needed per Investigator.
Period: Overall Study
Arm/Group | Stem Cell Collection Without In-vivo Purging With Bortezomib | Stem Cell Collection With In-vivo Purging With Bortezomib
Started | 51 | 50
Completed | 51 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stem Cell Collection Without In-vivo Purging With Bortezomib | Stem Cell Collection With In-vivo Purging With Bortezomib | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 29 | 66
  >=65 years | 14 | 21 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 49 | 46 | 95
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Multiparametric Flow Cytometry - Minimum Residual Disease
Description: Estimate the proportion of subjects with plasma cell contamination (defined as >0.01% and at least 100 cellular events) of harvested stem cell product by multi parametric flow cytometry (MFC) from patients with myeloma undergoing autologous stem cell collection 1) by standard of care mobilization using Granulocyte colony-stimulating factor (G-CSF) with or without Mozobil and 2) after two doses of bortezomib as in vivo purging plus standard of care using G-CSF with or without Mozobil.
Time Frame: Day 0 for all subjects (Day 0 is the day of stem cell collection)
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Collection Without In-vivo Purging With Bortezomib | Stem Cell Collection With In-vivo Purging With Bortezomib
Number analyzed (Participants) | 51 | 50
Participants | 11 | 13

2. Secondary Outcome: Multiparametric Flow Cytometry - Cluster of Differentiation 34 (CD34)Assessment
Description: Estimate the proportion of subjects who have a successful collection of stem cells (> 2 million Cluster of Differentiation 34 (CD34) cells/Kg of body weight) for autologous transplant in both treatment groups.
Time Frame: Within the first 30 days after stem cell collection
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Collection Without In-vivo Purging With Bortezomib | Stem Cell Collection With In-vivo Purging With Bortezomib
Number analyzed (Participants) | 51 | 50
Participants | 51 | 50

3. Secondary Outcome: Cluster of Differentiation 34 (CD34) Enumeration
Description: Estimate the percentage of Cluster of Differentiation 34 (CD34) positive cells in circulating peripheral blood as a measure of mobilization on the days of collection.
Time Frame: Within the first 30 days after stem cell collection
Measure: Mean (Standard Deviation); unit: percentage of CD34 positive cells
Arm/Group | Stem Cell Collection Without In-vivo Purging With Bortezomib | Stem Cell Collection With In-vivo Purging With Bortezomib
Number analyzed (Participants) | 51 | 50
percentage of CD34 positive cells | 8.9 (0.1) | 7.8 (0.1)

ADVERSE EVENTS:
Time Frame: From the time of signing the consent until 30 days after collection or up to 2 months.
Arm/Group | Stem Cell Collection Without In-vivo Purging With Bortezomib | Stem Cell Collection With In-vivo Purging With Bortezomib
All-Cause Mortality (participants affected / at risk) | 3/51 | 1/50
Serious Adverse Events (participants affected / at risk) | 12/51 | 24/50
Other Adverse Events (participants affected / at risk) | 39/51 | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Collection Without In-vivo Purging With Bortezomib (N=51) | Stem Cell Collection With In-vivo Purging With Bortezomib (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (8) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Collection Without In-vivo Purging With Bortezomib (N=51) | Stem Cell Collection With In-vivo Purging With Bortezomib (N=50)
Anemia (Blood and lymphatic system disorders) | 9 (26) | 7 (8)
Anorexia (Metabolism and nutrition disorders) | 26 (34) | 27 (33)
Anxiety (Psychiatric disorders) | 11 (11) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 8 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (7)
Constipation (Gastrointestinal disorders) | 15 (16) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 29 (55) | 29 (45)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (7)
Edema limbs (General disorders) | 12 (14) | 10 (11)
Fatigue (General disorders) | 21 (32) | 21 (30)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 (12) | 15 (16)
Hypertension (Vascular disorders) | 9 (14) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 27 (53) | 19 (43)
Hypomagnesemia (Metabolism and nutrition disorders) | 14 (16) | 7 (13)
Hyponatremia (Metabolism and nutrition disorders) | 9 (16) | 7 (9)
Insomnia (Psychiatric disorders) | 13 (15) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 20 (27) | 18 (28)
Nausea (Gastrointestinal disorders) | 33 (59) | 29 (45)
Neutrophil count decreased (Investigations) | 21 (37) | 16 (24)
Platelet count decreased (Investigations) | 25 (68) | 18 (24)
Vomiting (Gastrointestinal disorders) | 24 (37) | 21 (27)
White blood cell decreased (Investigations) | 27 (46) | 23 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02703779/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT02703779/ICF_001.pdf